CLINICAL TRIAL: NCT05456477
Title: A Randomized, Crossover Trial to Assess the Effects of Diets Containing Lean Beef vs. White Meat on Pancreatic Beta-cell Function in Men and Women With Prediabetes
Brief Title: A Trial to Assess Diets Containing Beef vs. Poultry on Pancreatic Beta-Cell Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MB-2112
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State | interventions — Red Meat; Poultry

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Beef (Experimental): Subject will consume beef entrees each day of the study period, and will not consume any additional meat, poultry, seafood, and eggs, other than the study entrees.
  Interventions: Other: Beef
- Poultry (Active Comparator): Subject will consume poultry entrees each day of the study period, and will not consume any additional meat, poultry, seafood, and eggs, other than the study entrees.
  Interventions: Other: Poultry

INTERVENTIONS:
Other: Beef — Beef entrees
  Arms: Beef
Other: Poultry — Poultry entrees
  Arms: Poultry

SUMMARY:
The objective of this study is to assess and compare the effects of usual diets containing lean beef vs. lean poultry on pancreatic beta-cell responses in men and women with prediabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 74 y of age, inclusive.
2. Subject has a BMI of 25.0-39.9 kg/m2, inclusive.
3. Subject has a Vein Access Scale score of 7-10.
4. Subject has prediabetes as indicated by a fasting plasma glucose of 100-125 mg/dL and/or HbA1c of 5.7%-6.4% at screening.
5. Subject is normally active and judged by the Investigator to be in general good health on the basis of medical history and screening measurements.
6. Subject is willing to consume study-related foods and follow the dietary instructions during each 4-week treatment period.
7. Subject is willing to come to the clinic for study food pick-up if needed.
8. Subject is willing to follow his/her usual physical activity pattern throughout the study period.
9. Subject agrees to avoid meat, poultry, seafood, and eggs, other than the study entrées, for the duration of the treatment periods.
10. Subject has no plans to change smoking habits during the study period.
11. Subject is willing to refrain from consumption of recreational marijuana and alcoholic beverages for 24 h prior to each clinic visit.
12. Subject is willing to refrain from vigorous physical activity for 24 h prior to each clinic visit.
13. Subject is willing to abstain from tobacco/nicotine products and caffeine use for at least 1 h prior to and during each clinic visit.
14. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator and is willing to complete study procedures.

Exclusion Criteria:

1. Subject has a laboratory test result of clinical significance based on the judgment of the Principal Investigator or qualified designee.
2. Subject has fasting blood glucose ≥ 126 mg/dL and/or HbA1c ≥ 6.5% at screening and/or known type 1 or type 2 diabetes mellitus.
3. Subject has atherosclerotic cardiovascular disease including any of the following: clinical signs of atherosclerosis including peripheral arterial disease, abdominal aortic aneurysm, carotid artery disease (symptomatic [e.g., myocardial infarction, angina, transient ischemic attack, or stroke of carotid origin] or > 50% stenosis on angiography or ultrasound) or other forms of clinical atherosclerotic disease (e.g., renal artery disease).
4. Subject has history or presence of a clinically significant health condition that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
5. Subject has a history of cancer in the prior 2 years, other than non-melanoma skin cancer or carcinoma in situ of the cervix.
6. Subject has uncontrolled hypertension (systolic blood pressure ≥ 160 mm Hg and/or diastolic blood pressure ≥ 100 mm Hg) at screening.
7. Subject has unstable use (defined as initiation or change in dose) of anti-hypertensive medication or thyroid hormone replacement within 4 weeks of screening (Appendix 1).
8. Subject has used alpha- or beta-adrenergic blockers and/or high-dose (> 25 mg/d) thiazide diuretics within 4 weeks of screening (Appendix 1).
9. Subject has used diabetes medications including any alpha-glucosidase inhibitor, biguanide (metformin), thiazolidinedione, dipeptidyl peptidase-4 inhibitor, meglitinide, sulfonylurea, Sodium-glucose Cotransporter-2 inhibitor, or GLP-1 receptor agonist within 4 weeks of screening (Appendix 1).
10. Subject has used systemic corticosteroids within 4 weeks of screening (Appendix 1).
11. Subject has used weight-loss drugs (including over-the-counter medications and/or supplements) or programs within 4 weeks prior to screening (Appendix 1).
12. Subject has used dietary supplements that may affect carbohydrate metabolism, including chromium picolinate, ginseng, cinnamon (as a supplement) and starch blockers within 2 weeks of screening (Appendix 1).
13. Subject has used any lipid altering drug therapy except stable use statin therapy (stable use is defined as no change in agent, dose, or regimen in the 4 weeks prior to screening).
14. Subject has had a weight change of ± 4.5 kg (10 lbs) in the previous 3 months.
15. Subject has an active infection and/or is on antibiotic therapy. Subject can be rescheduled for screening at least 7 days after completion of antibiotic therapy.
16. Subject has restrictive dietary habits (e.g., vegan, vegetarian, or very low carbohydrate diet).
17. Subject has a history of a diagnosed eating disorder (e.g., anorexia or bulimia nervosa).
18. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
19. Subject has a known allergy, sensitivity, or intolerance to any of the study foods.
20. Subject has been exposed to any non-registered drug product within 30 days of screening.
21. Subject has a current or recent history (past 12 months of screening) or strong potential for illicit drug or alcohol abuse. Alcohol abuse will be defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
22. Subject has a condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Ratio of incremental area under the curve (iAUC) for C-peptide to iAUC for glucose | 4 weeks

SECONDARY OUTCOMES:
Insulin sensitivity | 4 weeks
  The percent change during each treatment period in the Matsuda index where insulin resistance is defined as a value on the matsuda index of less than 3.
Fasting C-peptide | 4 weeks
  Change or percent change from baseline to the end of treatment of fasting C-peptide.
Insulin | 4 weeks
  Change or percent change from baseline to the end of treatment of insulin.
Mixed meal tolerance test (MTT) Disposition index | 4 weeks
  Change or percent change from baseline to the end of treatment of mixed meal tolerance test (MTT) disposition index.
Homeostasis model assessments of pancreatic beta-cell function (HOMA2%B) | 4 weeks
  Change or percent change from baseline to the end of treatment of homeostasis model assessment of pancreatic beta-cell function (HOMA2%B).
Homeostasis model assessments of insulin sensitivity (HOMA2%S) | 4 weeks
  Change or percent change from baseline to the end of treatment of homeostasis model assessment of insulin sensitivity (HOMA2%S).
Glucagon | 4 weeks
  Total AUC and iAUC for glucagon.
Glucagon-like petide-1 (GLP-1) | 4 weeks
  Total AUC and iAUC for glucagon-like peptide-1.
Glucose-dependent inhibitory polypeptide (GIP) | 4 weeks
  Total AUC and iAUC for glucose-dependent inhibitory polypeptide.
High-sensitivity C-reactive protein | 4 weeks
  Changes or percent changes from baseline to the end of treatment
Fibrinogen | 4 weeks
  Changes or percent changes from baseline to the end of treatment
Tumor necrosis factor alpha | 4 weeks
  Changes or percent changes from baseline to the end of treatment
Interleukin-6 | 4 weeks
  Changes or percent changes from baseline to the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Study Director — MB Clinical Research & Consulting, LLC
Locations (1):
- Illinois Institute of Technology, Chicago, Illinois, United States

REFERENCES:
- [Derived] Guzman E, Edirisinghe I, Wilcox ML, Kirkpatrick CF, Adams CG, Burton-Freeman BM, Maki KC. Effects of Diets Containing Beef Compared with Poultry on Pancreatic beta-Cell Function and Other Cardiometabolic Health Indicators in Males and Females with Prediabetes: A Randomized, Crossover Trial. Curr Dev Nutr. 2025 Oct 30;9(12):107589. doi: 10.1016/j.cdnut.2025.107589. eCollection 2025 Dec. PMID 41377490